CLINICAL TRIAL: NCT03362775
Title: EEG Analysis During Light Propofol Sedation
Acronym: MOTANA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Philippe GUERCI, M.D., PhD, ph, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PSS 2017/MOTANA-SCHMARTZ/MS
Record Dates: First submitted 2017-11-27; First posted 2017-12-05 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Electroencephalography
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Every subject will have an EEG recording in the absence of propofol, or during light sedation with propofol at an effect-site target concentration of 0.5 µg/mL and 1.0 µg/mL. Each subject will be his own control.
Masking Description: EEG will be electronically recorded and anonymised. The outcome assessor will analyse the EEG without knowledge of the propofol concentration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All subjects (Other): EEG will be recorded in all subjects before (0.0 µL/mL) and during a target controlled infusion of propofol (0.5 µL/mL and 1.0 µL/mL).
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Target-controlled infusion of propofol with an effect-site concentration of 0.0 µL/mL; 0.5 µL/mL and 1.0 µL/mL.

SUMMARY:
The hypothesis of this study is that propofol sedation does not affect the detectability of a movement intention in the EEG motor cortex signal. EEG signals will be recorded during the realization of intentional movements and movement intentions by the healthy volunteers, as well as during median nerve stimulation before and during propofol perfusion according to a target control infusion. (0 µg/mL; 0.5 µg/mL and 1 µg/mL).

DETAILED DESCRIPTION:
During an anesthesia, 0.1 to 0.2% of patients have an unexpected per-operative awakening, with the risk to have serious psychological consequences.

During a per-operative awakening, one of the first reflex of the patient is to move, but this is often not possible due to the use of neuromuscular blocking agents during the surgical procedure.

It is possible to detect a movement intention by analyzing the motor cortex EEG signal in awake volunteers. The same signal is present during light, non-painful median nerve stimulation.

The aim of this study is to determine wether this EEG signal can still be detected during light sedation by propofol, a drug commonly used during anesthesia. The investigators will include healthy male volunteers, who will make real movements, imagine a movement and have median nerve stimulations before and during a propofol infusion. The propofol will be infused according to a target controlled infusion with a effect-site concentration of 0.5 µg/mL and 1.0 µg/mL. Primary outcome is the detectability of event related desynchronization and event related synchronization in the EEG signal in the presence of propofol compared to the recordings without propofol

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Male
* affiliated to French social security
* normal physical examination
* 22 < body mass index < 28

Exclusion Criteria:

* Female
* allergy to propofol or one of the emulsion compounds (soja, egg)
* any pathology which may influence EEG recording or nerve conduction, such as diabetes, neuropathy, epilepsy, depression, psychotropic drug usage, drug usage)
* any allergic reaction associated with anesthesia

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ERD/ERS amplitude | 2 hours, during the experimentation
  Amplitude of event-related synchronization (ERS) and event-related desynchronization (ERD) will be recorded within 2 seconds of each motor task (real movement, imaginary movement) as well as median nerve stimulation. This amplitude will be compared tio the value recorded in the absence of propofol.

SECONDARY OUTCOMES:
Dose relationship between ERD/ERS and propofol concentration | 2 hours, during the experimentation
  Investigators will analyze wether there is a relationship between the propofol concentration and the ERD/ERS.
Detection ERS after median nerve stimulation | 2 hours, during the experimentation
  Investigators will test wether an ERS is present during propofol infusion at the effect-site concentrations of 0.5 µL/ml and 1.0 µL/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Rimbert, Study Chair — Institut National de Recherche en Informatique et en Automatique; Philippe GUERCI, MD, Principal Investigator — CHRU de NANCY
Locations (1):
- Department of Anesthesiology and Critical Care Medicine - University Hospital of Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blokland YM, Farquhar JD, Mourisse J, Scheffer GJ, Lerou JG, Bruhn J. Towards a novel monitor of intraoperative awareness: selecting paradigm settings for a movement-based brain-computer interface. PLoS One. 2012;7(9):e44336. doi: 10.1371/journal.pone.0044336. Epub 2012 Sep 6. PMID 22970202
- [Background] Blokland Y, Farquhar J, Lerou J, Mourisse J, Scheffer GJ, Geffen GJ, Spyrou L, Bruhn J. Decoding motor responses from the EEG during altered states of consciousness induced by propofol. J Neural Eng. 2016 Apr;13(2):026014. doi: 10.1088/1741-2560/13/2/026014. Epub 2016 Feb 9. PMID 26859192
- [Background] Lindig-Leon C, Bougrain L. Comparison of sensorimotor rhythms in EEG signals during simple and combined motor imageries over the contra and ipsilateral hemispheres. Annu Int Conf IEEE Eng Med Biol Soc. 2015;2015:3953-6. doi: 10.1109/EMBC.2015.7319259. PMID 26737159
- [Derived] Rimbert S, Schmartz D, Bougrain L, Meistelman C, Baumann C, Guerci P. MOTANA: study protocol to investigate motor cerebral activity during a propofol sedation. Trials. 2019 Aug 28;20(1):534. doi: 10.1186/s13063-019-3596-9. PMID 31455386